CLINICAL TRIAL: NCT05352542
Title: A Phase I Clinical Trial for Evaluating the Safety, Tolerance and Efficacy of GPC3-targeting CART Cell in Treatment of Advanced Hepatocellular Carcinoma
Brief Title: GPC3-targeting CART Cell in Treatment of Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: achieve the proof of concept
Sponsor: jianming xu (Other)
Responsible Party: Sponsor-Investigator, jianming xu, Leading Site Principal Investigator, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Organization: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPC3-targeting Study
Record Dates: First submitted 2022-04-01; First posted 2022-04-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPC3 Targeting CART Cells (Experimental): Each subject will receive GPC3 Targeting CART cells
  Interventions: Biological: GPC3 Targeting CART Cells

INTERVENTIONS:
Biological: GPC3 Targeting CART Cells — before treatment with GPC3 Targeting CART cells, subjects will receive a conditioning regimen

SUMMARY:
A Phase I Clinical Trial for Evaluating the Safety, Tolerance and Efficacy of GPC3-targeting CART Cell in Treatment of Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
This is an open-label, dose escalation/expansion study to assess the safety, tolerability, and efficacy of CART cell in patients ≥ 18 years of age with relapsed or refractory advanced hepatocellular carcinoma. Patients who meet the eligibility criteria will receive cell infusion. The study will include the following sequential phases: screening, pre-treatment (cell product preparation; lymphodepleting chemotherapy), treatment and follow up

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have fully understood the possible risks and benefits of participating in this study, are willing to follow and able to complete all trial procedures, and have signed informed consent;
2. Age 18-75 years;
3. Patients diagnosed as advanced hepatocellular carcinoma (HCC) histopathologically or cytologically; Progression or intolerance after previous standard systemic therapy;
4. GPC3 is detected positive by immunohistochemistry (IHC);
5. Child-Pugh score ≤ 7;
6. At least one assessable tumor lesion;
7. ECOG score: 0-1;
8. Expected survival ≥ 3 months;
9. Clinical laboratory values meet screening visit criteria

Exclusion Criteria:

1. Previous CAR-T cell, TCR-T cell or other cell therapies or therapeutic tumor vaccination directed at any target;
2. Any previous GPC3 targeted therapy;
3. Prior antitumor therapy with insufficient washout period;
4. Brain metastases with central nervous system symptoms;
5. Pregnant or lactating women
6. HCV-Ab or/and HIV-Ab positive; active syphilis;
7. Severe underlying diseases
8. Any condition that, in the opinion of the investigator, will make the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 2 years after CART infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment
Dose-limiting toxicity (DLT) rate | Minimum 2 years after CART infusion (Day 1)
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.
Recommended Phase 2 dose (RP2D) finding | 30 days after CART infusion (Day 1)
  RP2D established through ATD+BOIN design
CAR positive T cells | Minimum 2 years after CART infusion (Day 1)
  CAR positive T cells after CART infusion
CAR transgene levels in peripheral blood | Minimum 2 years after CART infusion (Day 1)
  CAR transgene levels in peripheral blood after CART infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | Minimum 2 years after CART infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via CART cell infusion, and the objective tumor response rate will be calculated for patients with measurable disease per RECIST 1.1 only
Disease control rate (DCR) | Minimum 2 years after CART infusion (Day 1)
  Disease Control Rate (DCR) is defined as the proportion of patients with complete response, partial responses and stable disease
Duration of Response(DoR) | Minimum 2 years after CART infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (according to RECIST 1.1) of the responders (who achieve PR or better response)
Time to Response (TTR) | Minimum 2 years after CART infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of CART to the date of the first response evaluation of the subject who has met all criteria for PR or better
Progress Free Survival (PFS) | 2 years after CART infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the CART to the first documented disease progression (according to RECIST 1.1) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Minimum 2 years after CART infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of CART to death of the subject
Incidence of anti-CART antibody | Minimum 2 years after CART infusion (Day 1)
  Venous blood samples will be collected to measure CART positive cell concentrations and the transgenic level of CART, at the time points when anti-CART antibody serum samples are evaluated

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gobroad Boren Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No